CLINICAL TRIAL: NCT02521857
Title: A Phase 1 Study to Evaluate the Impact of Water Consumption on the Pharmacokinetics of Sublingually Administered ALKS 5461
Brief Title: A Water Consumption Study of ALKS 5461 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK5461-A110
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Alkermes; Samidorphan; ALKS 5461; Healthy Volunteer; Pharmacokinetics
MeSH Terms: interventions — ALKS 5461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALKS 5461 (Experimental): Sublingual tablet
  Interventions: Drug: ALKS 5461

INTERVENTIONS:
Drug: ALKS 5461 — Sublingual tablet administered followed by consumption of 240 mL (8 ounces) of water at different timepoints

SUMMARY:
This study will evaluate the impact of water consumption on the pharmacokinetics of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) of 18.0 - 30.0 kg/m^2
* Is in good physical health
* Agrees to use an approved method of contraception for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Is currently pregnant or breastfeeding
* Has a history of substance abuse disorder
* Has used nicotine within 90 days prior to the study or anticipates a need to use nicotine during the study period
* Has used any prescription or over-the-counter medication, including natural health products or dietary supplements (with the exception of prescription contraceptives or hormonal replacements, acetaminophen, ibuprofen, or multivitamins) within 14 days prior to study start
* Has used opioids within 30 days prior to screening, or has an anticipated need for opioid medication at any point during the study
* Has used alcohol within 72 hours prior to any inpatient period
* Is a heavy caffeine drinker (regularly consuming 5 or more caffeinated beverages per day)
* Has a history of intolerance or hypersensitivity to opioids (buprenorphine) or opioid antagonists (naltrexone, naloxone)
* Additional criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
AUCinf | Up to 72 hours
  Area under the plasma concentration-time curve from time 0 to infinity for ALKS 5461
AUClast | Up to 72 hours
  Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration for ALKS 5461
Cmax | Up to 72 hours
  Maximum observed plasma concentration for ALKS 5461

SECONDARY OUTCOMES:
Safety and tolerability will be measured by the incidence of Adverse Effects | Up to 46 days

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Stanford, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigational Site, Overland Park, Kansas, United States